CLINICAL TRIAL: NCT04493112
Title: SeQuent Please Neo Multicenter Registry / Registro Multicéntrico Sequent Please NEO
Brief Title: SeQuent Please Neo Multicenter Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sequent Please NEO
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Drug Coating Balloon (DCB), Sequent Please
Keywords: Drug coating Balloon (DCB), Sequent Please
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry evaluates the safety and efficacy of paclitaxel-releasing SeQuent® Please Neo balloon in the following scenarios: restenosis, bifurcation lesions, small vessel lesions, diabetes (diffuse disease) and atrial fibrillation. The objective is to determine the success of the procedure and the preservation of vascular permeability.

DETAILED DESCRIPTION:
The preset registry aim is to evaluate the safety and efficacy of paclitaxel-releasing SeQuent® Please Neo balloon in the following scenarios: restenosis, bifurcation lesions, small vessel lesions, diabetes (diffuse disease) and atrial fibrillation. The principal objective is to determine the success of the procedure and the preservation of vascular permeability.

ELIGIBILITY:
Inclusion Criteria:

* ISR in a coronary artery with a diameter stenosis of at least 70%, a length of the stented segment of <25 mm, and a vascular diameter of at least 2.5 and up to 3.5 mm

Exclusion Criteria:

* There is no exclusion criteria except those patients with contraindication for antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 patients approx per site who fulfill inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Revascularization (TLR) with clinical follow-up at 12 months. | From baseline to 12 months
  Target Lesion Revascularization (TLR) with clinical follow-up at 12 months.

SECONDARY OUTCOMES:
Success of balloon dilation. | Baseline
  Success of balloon dilation.
Acute adverse cardiac events rate (MACE) and and MACE rate accumulated at 12 months. | From baseline to 12 months
  MACE rate and MACE rate accumulated at 12 months.
Premature follow-up indication | From baseline to 12 months
  Premature follow-up indication

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Rodriguez, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain